CLINICAL TRIAL: NCT06199648
Title: Digital Solutions for Elderly Care by Informal Caregivers: A Study on Nursing Benefits
Brief Title: Digital Solutions for Elderly Care by Informal Caregivers
Acronym: DigiSECC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences for Health Professions Upper Austria (Other)
Collaborators: LICA Life Care GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: DigiSecc 001
Record Dates: First submitted 2023-11-21; First posted 2024-01-10 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Activities of Daily Living
Keywords: Caregivers*; Frail Elderly*; Humans; Austria; Telemedicine
MeSH Terms: interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only pseudonymous, blinded data will be provided to statisticians for analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: web-based documentation and advice (Experimental)
  Interventions: Other: web-based documentation and advice
- Arm B: Standard of care (No Intervention)

INTERVENTIONS:
Other: web-based documentation and advice — Caregivers will be supported with a web-based documentation and advice system for home care for elderly people
  Arms: Arm A: web-based documentation and advice

SUMMARY:
The study aims to determine the benefits of a web-based documentation and advice for elderly people and their caregivers. It is a randomized controlled trial with two arms (intervention, control). While the participants will be supported by a web-based application within the intervention, they will receive standard care only in the control. In addition, a follow-up until the end of the study will be realized.

DETAILED DESCRIPTION:
Background: The majority of elderly people want to live at home, and the home care they need is often provided by informal caregivers. In addition, the number of elderly people is increasing while the number of people who can support them is decreasing. It is therefore important to improve the quality of care and support caregivers. Unfortunately, caregivers are often under heavy strain and the amount of time they can spend receiving advice and support is very limited. Web-based applications could be a solution to address the time needs of caregivers, but little is known about whether such applications are of benefit to the elderly themselves or their caregivers.

Description of the Intervention: A web-based documentation and advice application for home care for elderly people. The intervention is based on the daily status diary, the completion of daily tasks, the writing of short reports (if applicable) and the documentation of the caregiver's constitution. Adherence to the purpose of the web-based application is defined as entering data at least 5 out of 7 days per week.

It is a single-center, open-label, randomized controlled trial with two arms (intervention, control). The study consists of one in person screening visit, two in person study visits and 3 monthly follow-up visits via phone (Visit 0: Screening Visit, Visit 1: Baseline Visit, Visit 2: End of Study Visit, Visit 3: Follow-up). The study-related measurements are: Barthel Index, Short Form of the Late Life Function and Disability Instrument, 5-level EuroQol quality of life questionnaire (EQ-5D-5L), De Morton Mobility Index (DEMMI), individual's general self-efficacy (GSE), user experience questionnaire short form (UEQ-S), Adherence (minimum frequency with which the daily diary was completed by the caregiver). The study begins when both parties in the pair (elderly person and caregiver) sign the informed consent form and ends when the older person dies or the study ends, whichever comes first. The intervention period is 12 weeks.

ELIGIBILITY:
Key Inclusion Criteria for the Elderly Person:

* 55 years and older
* Community-dwelling
* Resident in Upper Austria
* Barthel Index below 100
* Requires assistance with activities of daily living

Key Exclusion Criteria for the Elderly Person:

* Planned nursing home admission in the next 12 weeks
* Chronic obstructive pulmonary disease stage III or IV
* Insufficient understanding and judgment to consent to the study

Main Inclusion Criteria for the Caregiver:

* Caregiver of an older person
* Tech savvy
* Committed to using an app to support caregiving

Main Exclusion Criteria for the Caregiver:

* 17 years and younger
* Insufficient insight and judgment to consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Mean change in function and disability of the elderly participant estimated with Barthel Index (BI) | 104 Weeks
  The BI assesses the functional status and independence in basic activities of daily living (ADL) of elderly people. Each domain is scored on a 0-5 or 0-10 scale, with the overall score ranging from 0 to 100. A higher score represents a higher level of independence. The BI will be rated by the study staff. The Hamburg Classification Manual provides detailed criteria for scoring.

SECONDARY OUTCOMES:
Mean change in function and disability of the elderly participant estimated with Short Form of the Late-Life Function and Disability Instrument (SF-LLFDI) | 104 Weeks
  The SF-LLFDI assesses two domains: function and disability, with various subdomains. It is a self-administered questionnaire that can be completed online or on paper, consisting of 32 items rated on a 5-point Likert scale. The scores are converted into a percentage of the maximum possible score for each subdomain and domain, with higher scores indicating better function or less disability. The SF-LLFDI will be self-rated by the elderly participant.
Mean change in quality of life of the elderly participant estimated using the 5-item and 5-dimension versions of the EuroQoL questionnaire (EQ-5D-5L) | 104 Weeks
  The EQ-5D-5L is a patient-reported outcome measure that assesses five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate their health status by ticking the box next to the most appropriate statement in each of the five dimensions. This results in a 5-digit number describing the patient's health. The EQ-5D-5L is self-reported by the elderly participant.
Mean change in mobility of the elderly participant estimated with the de Morton Mobility Index (DEMMI) | 104 Weeks
  The DEMMI is an advanced instrument designed to measure and monitor changes in mobility for older adults. It assesses tasks ranging from bed/bedside to dynamic balance and increases in difficulty. Each task is scored in each category 0, 1, or 2. The raw score maximum total is 19, and the converted score maximum total is 100. The DEMMI will be rated by a health professional.
Mean change in self-efficacy of the elderly participant estimated using the General Self-Efficacy Short Scale (GSE) | 104 Weeks
  The GSE measures general self-efficacy, which describes an individual's overall confidence in their own competence. It consists of ten items scored on a 4-point Likert-type scale. The total score ranges from 10 to 40, with higher scores indicating higher levels of general self-efficacy. The GSE is self-reported by the elderly participant.
Mean change in quality of life of the caregiver estimated with EQ-5D-5L | 104 Weeks
  The EQ-5D-5L is a patient-reported outcome measure that assesses five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his or her health status by ticking the box next to the most appropriate statement in each of the five dimensions. This results in a 5-digit number describing the patient's health. The EQ-5D-5L is self-reported by the caregiver.
User experience estimated with the UEQ-S | 1 Hour
  The UEQ-S measures the overall attractiveness of the web-based application in two domains of user experience: pragmatic quality and hedonic quality. Pragmatic quality refers to the usability, efficiency and clarity of the web-based application, while hedonic quality refers to the stimulation, interest and novelty of the web-based application. The UEQ-S is rated by the caregiver.
Change in status of the caregiver over time estimated with the daily caregiver status diary | 12 Weeks
  Caregivers rate their experience, effort and positive moments on a daily smiley scale of 1 to 5, with more smileys indicating a better rating. The data is exported for analysis and is also used to record adverse events related to the elderly person.
Adherence by days with no entry in the daily status diary | 12 Weeks
  Adherence is defined as the degree to which an individual uses an eHealth technology in accordance with the manufacturer's recommendations. In this study, adherence to the use of the application is assessed by examining the data entered by the caregiver into the daily status diary and the days with no entries. Adherence is defined as making entries on at least 5 days within a week in 9 out of 12 weeks (i.e. 75%).
Survival of the elderly participant based on the number of Grade 5 adverse events in the elderly participant estimated using an adverse event (AE) reporting form. | 104 Weeks
  Survival based on the number of Grade 5 adverse events experienced by the older participant, as recorded on an AE reporting form. A higher number of grade 5 adverse events indicates a lower survival rate.
Hospitalization rate, with the number of adverse events requiring hospitalization of the elderly participant estimated using an adverse event (AE) reporting form. | 104 Weeks
  The hospitalization rate is determined based on the number of adverse events requiring hospitalization experienced by the older participant, as recorded on an AE reporting form. A higher number of AEs reporting hospitalization indicates a higher hospitalization rate.
Safety, with number of adverse events estimated using an adverse event (AE) reporting form. | 104 Weeks
  Safety is determined by the number of adverse events experienced by the elderly participant and recorded on an AE reporting form. A higher number of adverse events indicates a lower level of safety.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mittermaier, Dr., Principal Investigator — Institute of Physical Medicine and Rehabilitation, Kepler University Hospital, Linz, Austria; Bernhard Schwartz, Dr. BSc MSc, Study Director — University of Applied Sciences for Health Professions Upper Austria
Locations (1):
- University of Applied Sciences for Health Professions Upper Austria, Linz, Upper Austria, Austria

IPD SHARING:
Plan to Share IPD: No